CLINICAL TRIAL: NCT05775848
Title: A Phase 3 Randomized, Placebo-controlled, Double-blind Study to Evaluate the Efficacy and Safety of BBP-418 (Ribitol) in Patients With Limb Girdle Muscular Dystrophy 2I (LGMD2I)
Brief Title: Study to Evaluate the Efficacy and Safety of BBP-418 (Ribitol) in Patients With Limb Girdle Muscular Dystrophy 2I (LGMD2I)
Acronym: Fortify
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ML Bio Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLB-01-005
Record Dates: First submitted 2023-02-16; First posted 2023-03-20 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Limb-Girdle Muscular Dystrophy Type 2I (LGMD2I)
MeSH Terms: conditions — Muscular Dystrophy, Limb-Girdle, Type 2I | interventions — Ribitol

STUDY DESIGN:
Intervention Model Description: Randomization will be stratified by mutation status (L276I homozygous or other), age (<12 years [to allow for possible addition of this age group in a future protocol amendment], 12 to <18 years, and 18 to 60 years of age), and qualification status for the Primary Efficacy Analysis Population ("qualifies" or "does not qualify").
  [NOTE: EU region will only enroll 18 to 60 years of age]
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 2:1 Randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BBP-418 (Active Comparator): BBP-418 Granules for Oral Solution will be supplied as granules in tri-ply PET/Aluminum/PE sachets for unit dose. The number of sachets to reconstitute will depend on the applicable dose to be delivered, 9 g BID or 12 g BID, as determined by the weight of the participant. The granules will be reconstituted in water for oral administration.
  Interventions: Drug: BBP-418 (ribitol); Other: Placebo
- Placebo to Match BBP-418 (Placebo Comparator): The placebo will be identical to the BBP-418 Granules for Oral Solution in appearance, packaging, labeling, and storage conditions.
  Interventions: Drug: BBP-418 (ribitol); Other: Placebo

INTERVENTIONS:
Drug: BBP-418 (ribitol) — The BBP-418 drug product is provided as Granules for Oral solution consisting of BBP-418 drug substance and silicon dioxide in a multilaminate sachet with a foil barrier. Silicon dioxide is generally regarded as safe and listed in the FDA IIAD. Silicon dioxide is a compendial excipient and is commonly used in pharmaceutical dosage forms. The BBP-418 Granules for Oral Solution are provided in sachets.The BBP-418 Granules for Oral Solution are reconstituted in water for oral administration.
Other: Placebo — A placebo matched for similar taste and appearance was compounded at the clinical pharmacy with sucralose as a 0.35 mg/mL oral solution in purified water (USP) in a glass container. Sucralose is similar in taste to the compounded drug product.

SUMMARY:
This study will evaluate the safety and efficacy of long-term administration of BBP-418 in patients with LGMD2I/R9. The study will include patients ages 12 to 60, consistent with the existing preclinical toxicology profile. This will encompass the significant majority of existing diagnosed patients based upon the established epidemiology of the disease.

ELIGIBILITY:
Participants must meet all the following criteria to be enrolled:

1. Have a genetically confirmed diagnosis of LGMD2I/R9 (including review of records of previous molecular genetic testing) and be clinically affected (defined as demonstrating clinical weakness on bedside evaluation in either a limb-girdle pattern, or in a distal extremity).
2. Male or female participants 12 to 60 years of age (inclusive). [NOTE: EU region will only enroll 18 to 60 years of age]
3. Have a body weight >30 kg.
4. The participant (or parent/guardian) who signs the ICF understands the study procedures and the participant agrees to participate in the study by giving informed consent (and assent, if <18 years of age).
5. Female participants of childbearing potential and male participants of reproductive potential must be willing to use a highly effective method of contraception from time of consent through 12 weeks after last dose.
6. Willing and able to complete all study procedures, including biopsies, according to the Schedule of Assessments (see Appendix 1).

Participants must not meet any of the following criteria to be enrolled:

1. Evidence of clinically significant concomitant disease, including:

   1. Any significant concomitant medical condition, including mental, cardiac, renal, pulmonary, hepatic, or endocrine disease other than that associated with LGMD2I/R9.
   2. Moderate to severe renal impairment (estimated glomerular filtration rate [eGFR] of < 60 mL/min/1.73 m2 based on cystatin C [CysC]), as calculated by the central laboratory.
   3. Any other laboratory, vital sign, ECG abnormality, clinical history, or finding that, in the Investigator's opinion, is likely to unfavorably alter the risk-benefit of study participation, confound study results, or interfere with study conduct or compliance.
   4. Surgery for scoliosis or other indication that will significantly impact the participant's ability to execute clinical assessments planned or expected to be required to manage curvature within 12 months following the Screening Visit.
2. A participant with a score of zero on any one or more of the primary or key secondary endpoints at the time of screening. (Participants who previously completed participation in Study MLB-01-001 and would be excluded due to this criterion may enroll in this study provided all inclusion and no other exclusion criteria are met.)
3. If pregnant and/or breastfeeding or planning to conceive children within the projected duration of the study through 12 weeks after the last dose of study treatment.
4. Use of ribose or other sugar alcohol-containing supplement within 90 days of the Screening Visit.
5. Use of a systemic corticosteroid for the treatment of muscular dystrophy within 90 days of the Screening Visit. (An inhaled corticosteroid or bronchodilator for reactive airway disease is allowed if the participant is on a stable dose for 30 days prior to study entry.)
6. Previously received gene therapy to treat LGMD2I/R9.
7. Participants with active suicidal ideation as measured by Columbia-Suicide Severity Rating Scale during screening with most severe suicide ideation score of 4 (Active Suicidal Ideation with Some Intent to Act, without Specific Plan) or 5 (Active Suicidal Ideation with Specific Plan and Intent).
8. Presence of a platelet disorder, bleeding disorder, or other contraindication to muscle biopsy.
9. Actively on an experimental therapy or device or was on an experimental therapy or device within 90 days of the Screening Visit, or was on BBP-418 at any time.
10. In the judgment of the Investigator or Medical Monitor, has any clinically important ongoing medical condition or laboratory abnormality or condition that might jeopardize the participant's safety, increase their risk from participation, or interfere with the study. For COVID-19 infections, Investigator should refer to local guidance.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in North Star Assessment for Limb Girdle Muscular Dystrophy following 36 months of treatment to assess efficacy of BBP-418 or placebo | 36 months
Frequency and severity of treatment-emergent adverse events following 36 months of treatment to assess safety of BBP-418 or placebo | 36 months

SECONDARY OUTCOMES:
Change from baseline in 10 meter walk test velocity to assess the clinical efficacy of BBP-418 in patients with LGMD2I/R9 | 36 months
Change from baseline in pulmonary function as measured by FVC (percent predicted, performed in a sitting position) to assess the clinical efficacy of BBP-418 in patients with LGMD2I/R9 | 36 months
Change from baseline in the Performance of Upper Limb scale 2.0 to assess the clinical efficacy of BBP-418 in patients with LGMD2I/R9 | 36 months

OTHER OUTCOMES:
Change from baseline in total glycosylated Alpha dystroglycan to assess biomarkers for clinical efficacy of BBP-418 in patients with LGMD2I/R9 | 36 months
Change from baseline in glycosylated Alpha dystroglycan / total glycosylated Alpha dystroglycan ratio to assess biomarkers for clinical efficacy of BBP-418 in patients with LGMD2I/R9 | 36 months

CONTACTS AND LOCATIONS:
Locations (21):
- United States (13):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California Irvine, Irvine, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Florida, Gainsville, Florida
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Minnesota, Twin Cities, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Oregon Health & Science University (OHSU) - Neurology Clinic - South Waterfront, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of the Kings Daughters, Norfolk, Virginia
- Royal Brisbane and Women's Hospital,, Brisbane, Queensland, Australia
- Rigshospitalet, Neuromuscular Clinic and Research Unit, Copenhagen, Denmark
- Charité Universitätsmedizin Berlin and Max Delbrück Center, Berlin, Germany
- IRCCS Ca' Granda Ospedale, Milan, Italy
- Leiden University Medical Center, Leiden, Netherlands
- Universitetssykehuset Nord-Norge, Department of Neurology, Tromsø, Norway
- United Kingdom (2):
  - Great Ormond Street Hospital for Children, London
  - International Centre for Life, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR